CLINICAL TRIAL: NCT00005089
Title: Evaluation of CHOP Plus Rituximab Plus Involved Field Radiotherapy for Stages I, IE, and Non-Bulky Stages II and IIE, CD20 Positive, High-Risk Localized Aggressive Histologies of Non-Hodgkin's Lymphoma
Brief Title: S0014 Combination Chemotherapy Plus Rituximab and Radiation Therapy in Treating Patients With Stage I or Stage II Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067707; S0014 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-04-06; First posted 2004-02-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; stage I adult Burkitt lymphoma; stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHOP + Rituximab + RT (Experimental): 3 21-day cycles of CHOP (cyclophosphamide 750 mg/m^2, doxorubicin 50 mg/m^2, vincristine 1.4 mg/m^2, prednisone 100 mg x 5 days) + Rituximab 375 mg/m^2 (x 2 days for cycle 1, x 3 days for cycles 2-3). RT 4000-5500 cGy given in 25 fractions starting 3 weeks after completion of CHOP + Rituximab.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: rituximab — 375 mg/m^2 on days 1,8 of cycle 1, then on days 1-3 of cycles 2-3.
Drug: cyclophosphamide — 750 mg/m^2 on day 10 of cycle 1, then on day 21 of cycles 2-3.
Drug: doxorubicin hydrochloride — 50 mg/m^2 on day 10 of cycle 1, then on day 21 of cycles 2-3.
Drug: prednisone — 100 mg on days 10-14 of cycle 1, then on days 3-7 of cycles 2-3.
Drug: vincristine sulfate — 1.4 mg/m^2 on day 10 of cycle 1, then on day 3 of cycles 2-3.
Radiation: radiation therapy — 4000-5500 cGy given in 25 fractions starting 3 weeks after completion of CHOP + Rituximab.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with monoclonal antibody therapy and radiation therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus rituximab and radiation therapy in treating patients who have stage I or stage II non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess two year progression free survival after treatment with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) plus rituximab followed by radiotherapy in patients with stage I, IE, or non-bulky stage II or IIE high risk localized intermediate or high grade non-Hodgkin's lymphoma. II. Determine the toxicity of this treatment in these patients.

OUTLINE: Patients receive rituximab IV on days 1 and 8 of the first course, then on day 1 of courses 2 and 3. Patients receive cyclophosphamide IV over 1-2 hours, doxorubicin IV, and vincristine IV on day 10 of the first course, then on day 3 of courses 2 and 3. Patients receive oral prednisone on days 10-14 of the first course, then on days 3-7 of courses 2 and 3. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Chemotherapy is followed by radiotherapy administered 5 days a week for 4-5 weeks. Patients are followed every 6 months for two years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage I, IE, or non-bulky II or IIE non-Hodgkin's lymphoma of one of the following subtypes: Diffuse large B-cell Mantle cell High grade B-cell, Burkitt's or Burkitt like Anaplastic large cell (B-cell phenotype only) Lymphoma must express CD20 All disease must be encompassable in a single radiation port (including any resected disease) Must have at least 1 of the following adverse prognostic features: Non-bulky stage II or non-bulky stage IIE disease Over 60 years of age Zubrod performance status of 2 Elevated serum LDH A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No medical contraindications to CHOP chemotherapy or rituximab No prior malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No AIDS or HIV Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior monoclonal antibody therapy Chemotherapy: No prior chemotherapy for lymphoma Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for lymphoma Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2000-04; Primary Completion 2004-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 6 weeks while on protocol treatment, then every 6 months for 2 years, then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Miller, MD, Study Chair — University of Arizona
Locations (92):
- United States (92):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Persky DO, Unger JM, Spier CM, Stea B, LeBlanc M, McCarty MJ, Rimsza LM, Fisher RI, Miller TP; Southwest Oncology Group. Phase II study of rituximab plus three cycles of CHOP and involved-field radiotherapy for patients with limited-stage aggressive B-cell lymphoma: Southwest Oncology Group study 0014. J Clin Oncol. 2008 May 10;26(14):2258-63. doi: 10.1200/JCO.2007.13.6929. Epub 2008 Apr 14. PMID 18413640
- [Result] Miller TP, Unger JM, Spier C, et al.: Effect of adding rituximab to three cycles of CHOP plus involved-field radiotherapy for limited-stage aggressive diffuse B-cell lymphoma (SWOG-0014). [Abstract] Blood 104 (11): A-158, 2004.
- [Derived] Stephens DM, Li H, LeBlanc ML, Puvvada SD, Persky D, Friedberg JW, Smith SM. Continued Risk of Relapse Independent of Treatment Modality in Limited-Stage Diffuse Large B-Cell Lymphoma: Final and Long-Term Analysis of Southwest Oncology Group Study S8736. J Clin Oncol. 2016 Sep 1;34(25):2997-3004. doi: 10.1200/JCO.2015.65.4582. Epub 2016 Jul 5. PMID 27382104